CLINICAL TRIAL: NCT06992960
Title: A Prospective, Randomised, Split-Body, Controlled, Non-Inferiority Clinical Study on the Scar Healing Effects of ChitoCare Medical Scar Healing Gel in Women Undergoing Breast Reduction or Mastopexy Surgery (CHITOSCAR)
Brief Title: Evaluation of the Scar Healing Effects of ChitoCare Medical Scar Healing Gel in Women Undergoing Breast Reduction or Mastopexy Surgery (CHITOSCAR)
Acronym: CHITOSCAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Primex ehf (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHITOSCAR-25-01
Record Dates: First submitted 2025-05-13; First posted 2025-05-28 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Surgical Scars

STUDY DESIGN:
Masking Description: Due to the nature of the trial, both the participants and investigators will know which treatment is which, however, photographs of scars will be assessed by a blinded evaluator once all data collection is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): ChitoCare® medical Scar Healing Gel (Örsáragel) administered topically twice daily for 6 months post-surgery
  Interventions: Device: ChitoCare® medical Scar Healing Gel (Örsáragel)
- Control (Active Comparator): Amoena CuraScar Mammilla Circles Silicone Scar Patch and Amoena CuraScar Anchors Silicone Scar Patch worn daily (continuous use, minimum 12 hrs per day as per the IFU) for 6 months post-surgery
  Interventions: Device: Amoena CuraScar Mammilla Circles Silicone Scar Patch and Amoena CuraScar Anchors Silicone Scar Patch

INTERVENTIONS:
Device: ChitoCare® medical Scar Healing Gel (Örsáragel) — ChitoCare® medical Scar Healing Gel is a topical gel indicated for the treatment of new and old scars. The Scar Healing Gel provides a soothing effect and support to the scar tissue to heal in an orderly manner. It protects against infections, stimulates cell proliferation in old and new scars, as well as correct tissue organization with proper collagen alignment for a better aesthetic appearance and skin flexibility. Ideal for treating scars after accidents, surgery, C-section and cosmetic surgery. For smoother and less visible scars. May be used by the whole population, also elderly and children.
  Arms: Active
Device: Amoena CuraScar Mammilla Circles Silicone Scar Patch and Amoena CuraScar Anchors Silicone Scar Patch — Amoena CuraScar Mammilla Circles Silicone Scar Patch and Amoena CuraScar Anchors Silicone Scar Patch are silicon-based, single-patient, multi-use scar patches intended for use as scar reduction therapy in surgical breast scars. The silicone creates a moist environment on the scar, which prevents the scar from drying out. It keeps the scar soft and has a positive effect on scar tissue. The devices are specifically designed for breast scarring and are shaped to fit the normal surgical scars experienced after breast surgery.
  Arms: Control

SUMMARY:
Patients undergoing breast reduction or mastopexy surgery will be screened and recruited for participation in the study. Eligible patients will act as their own control with one breast receiving the active intervention (ChitoCare® medical Scar Healing Gel) and the other receiving standard of care (Amoena CuraScar Mammilla Circles Silicone Scar Patch and Amoena CuraScar Anchors Silicone Scar Patch). The active and control interventions will be applied for six months, and participants will be followed for up to 12 months. The scar properties of each breast will be assessed at study initiation (Day 0) and at study visits at 3, 6, 9, and 12 months using the Patient and Observer Scar Assessment Scale (POSAS) and via blinded assessment of photographs. Other subjective parameters such as pain, itching, and overall perception of the healed wound will be collected at each study visit via the POSAS, and patients' opinion, preferences, and compliance regarding the treatments will be collected via a basic questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be given
* Female ≥ 18 years old
* Having planned or very recently (within 21 days) undergone breast reduction or mastopexy surgery on both breasts
* Not yet begun any treatment aimed at reducing scarring
* Wound is not infected at the time of enrolment
* Able to understand and comply with the requirements of the study

Exclusion Criteria:

* Patients with serious concomitant disease (cancer, heart failure (NYHA class IV), severe anaemia (Hb<100 g/L), neoplasia)
* Any significant condition that may preclude the participant from the study (e.g. severe depression or psychiatric illness)
* Patients who will require additional surgical procedures during the study
* Patients diagnosed with autoimmune connective tissue diseases
* Previous treatment under this clinical protocol
* Participation in another clinical trial
* Receiving or scheduled to receive a medication or treatment which, in the opinion of the investigator, is known to interfere with, or affect the rate and quality of wound healing
* Allergy to shellfish* (if unknown, the patient may try a small sample of the IP on their intact skin to assess for any potential allergic reaction.)
* Medical condition likely to require systemic corticosteroids during the study period
* Pregnant or lactating women
* Smoker

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 39 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Comparison of scar assessment at 12 months | 12 months post-surgery
  Comparison of the subjective assessment of scar appearance using the Patient and Observer Scar Assessment Scale 3.0 (POSAS) in active vs control group at 12-months post-surgery.
  The POSAS 3.0, for both the Patient Scale and the Observer Scale, rates each individual item on a 5-point scale.
  The minimum value for an item is 1, which corresponds to a scar characteristic or sensation that is like normal skin (a better outcome). The maximum value for an item is 5, which indicates the largest difference from normal skin or the worst imaginable scar characteristic or sensation (a worse outcome).
  The total score for the Patient Scale and the Observer Scale is calculated by summing the scores of the individual items within each scale. Consequently, for the POSAS 3.0, a higher total score on either the Patient Scale or the Observer Scale signifies a worse scar outcome or a greater severity of scar-related issues from that perspective.

SECONDARY OUTCOMES:
Comparison of scar assessment at 3, 6, and 9 months | 3, 6, and 9 months post-surgery
  Comparison of the subjective assessment of scar appearance using the Patient and Observer Scar Assessment Scale (POSAS) in active vs control group at 3, 6, and 9 months post-surgery.
  The POSAS 3.0, for both the Patient Scale and the Observer Scale, rates each individual item on a 5-point scale.
  The minimum value for an item is 1, which corresponds to a scar characteristic or sensation that is like normal skin (a better outcome). The maximum value for an item is 5, which indicates the largest difference from normal skin or the worst imaginable scar characteristic or sensation (a worse outcome).
  The total score for the Patient Scale and the Observer Scale is calculated by summing the scores of the individual items within each scale. Consequently, for the POSAS 3.0, a higher total score on either the Patient Scale or the Observer Scale signifies a worse scar outcome or a greater severity of scar-related issues from that perspective.
Improvement in subjective assessment of scar tissue | 3, 6, 9, and 12 months post-surgery
  Improvement of the subjective assessment of scar tissue between Day 0 and 3, 6, 9, and 12 months using the POSAS in active vs control arm.
  The POSAS 3.0, for both the Patient Scale and the Observer Scale, rates each individual item on a 5-point scale.
  The minimum value for an item is 1, which corresponds to a scar characteristic or sensation that is like normal skin (a better outcome). The maximum value for an item is 5, which indicates the largest difference from normal skin or the worst imaginable scar characteristic or sensation (a worse outcome).
  The total score for the Patient Scale and the Observer Scale is calculated by summing the scores of the individual items within each scale. Consequently, for the POSAS 3.0, a higher total score on either the Patient Scale or the Observer Scale signifies a worse scar outcome or a greater severity of scar-related issues from that perspective.
Blinded assessment of scars | 3, 6, 9, and 12 months post-surgery
  Comparison of scar appearance at 3, 6, 9, and 12 months as judged by blinded assessment of photographs of active vs control intervention using the modified Stony Brook Scar Evaluation Scale (mSBSES).
  For the modified SBSES, the scoring is structured such that higher scores indicate a better cosmetic outcome or less noticeable scarring. Scar width, height, colour, and presence of incision line are rated on a scale for 0-2, where 0 indicates a worse outcome, and 2 indicates similarity to normal skin. The best possible score is therefore 8, and worst outcome is 0.
Comparison of pain, discomfort, itching, and range of motion | 3, 6, 9, and 12 months post-surgery
  Comparison of pain or discomfort, itching, range of motion etc. between the groups as captured by the POSAS at 3, 6, 9, and 12 months.
  The POSAS 3.0, for both the Patient Scale and the Observer Scale, rates each individual item on a 5-point scale.
  The minimum value for an item is 1, which corresponds to a scar characteristic or sensation that is like normal skin (a better outcome). The maximum value for an item is 5, which indicates the largest difference from normal skin or the worst imaginable scar characteristic or sensation (a worse outcome).
  The total score for the Patient Scale and the Observer Scale is calculated by summing the scores of the individual items within each scale. Consequently, for the POSAS 3.0, a higher total score on either the Patient Scale or the Observer Scale signifies a worse scar outcome or a greater severity of scar-related issues from that perspective.
Adverse events | 12 months post-surgery
  Incidence of adverse events between arms
Comparison of treatment compliance | 6 months post-surgery
  Participants will be asked at 3 months and 6 months post-surgery how they would rate their compliance to each treatment (arm) via a basic questionnaire: a 5-point rating system will ask whether participants used/wore their treatment every day as recommended, most days but not always, only sometimes, rarely, or hardly ever/did no comply to treatment. Scores between the 2 arms will be compared for trends for treatment compliance.
Cost comparison of treatments | 6 months post-surgery
  Cost of active vs control treatment in relation to outcomes over 6 months
Patient treatment preference | 3 and 6 months post-surgery
  Participants will be asked which treatment they preferred (i.e., active vs control treatment) via a questionnaire at 3 and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Klíníkin Ármúla, Reykjavik, Capital Region, Iceland

IPD SHARING:
Plan to Share IPD: No